CLINICAL TRIAL: NCT03775720
Title: Does Disclosing Genetic Risk to Salt Sensitivity Increase Compliance to Personalised Dietary Recommendations?
Brief Title: Disclosure of Genetic Risk for Salt Sensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Principal Investigator, Kim Wright, Research Administrator, St Mary's University College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMEC_2017-18_142
Record Dates: First submitted 2018-09-21; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Salt-sensitive Hypertension
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low genetic risk group (Experimental): Dietary advice to maintain salt intake to 6g/day
  Interventions: Behavioral: Dietary advice
- High genetic risk group (Experimental): Dietary advice to reduce salt intake to 4g/day
  Interventions: Behavioral: Dietary advice

INTERVENTIONS:
Behavioral: Dietary advice — Based on their genetic risk, participants are given advice to either adhere to general dietary guidelines related to salt intake or to reduce their salt intake to no more than 4 grams per day.

SUMMARY:
The global burden of cardiovascular disease (CVD) has decreased over the past 10 years. Nevertheless, the disease still kills one in three people. Hypertension is one of the leading causes of cardiovascular disease, with salt in the diet being a main contributor. Depending on an individual's DNA, participants may or may not be salt sensitive. Genotyping individuals for variants in a salt sensitivity gene (SLC4A5) may identify salt sensitive individuals which may benefit from a personalised dietary advice to reduce salt intake. Adherence to such advice can then be assessed which may aid in prevention of hypertension and CVD.

DETAILED DESCRIPTION:
Salt sensitivity is a key risk factor for hypertension. However, population decrease in salt intake is less than optimal. Research suggests genetics-based personalised nutrition can positively impact health behaviours aiding in the prevention of chronic disease development. However, the effects of communicating such information are unclear. The aims of this study will be to analyse the impact of communicating genetic susceptibility to salt sensitivity on salt intake by assessing dietary salt intake before and after disclosure of genetic risk for hypertension according to the polymorphism in the SLC4A5. Participants will be normotensive, aged 18-35 years. All individuals will receive genetics-based personalised nutritional information. Participants displaying the risk genotype (AA + AC) will be advised to decrease salt intake to less than 4g/d and non-risk will be advised to adhere to government recommendations (6g/d). Dietary recall (24hrs) and 24-hour urine collection will be collected at baseline and four-weeks post-intervention to assess salt intake and excretion.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females, aged 18-35

Exclusion Criteria:

* pregnant, CVD events (Angina, myocardial infarction, heart failure) or stage 2, hypertension, a BMI ≥30kg/m2, or experiencing mental anguish.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Dietary salt intake | 1 month
  24-hour recall

IPD SHARING:
Plan to Share IPD: No